CLINICAL TRIAL: NCT04788329
Title: The Effect of Mindfulness Programs on Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-01495
Record Dates: First submitted 2021-03-05; First posted 2021-03-09 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Relaxation Group (Experimental): This program teaches patients how to feel calmer before surgery. Patients are taught relaxation techniques by phone or in person by trained NYU personnel.
  Interventions: Behavioral: "Prepare for Surgery, Heal Faster" Program
- Meditation Group (Experimental): This treatment group will be enrolled in Wim Hof Method, a meditation program. Patients in this group will take the online "The Fundamentals Course" provided by the Wim Hof Method. The patients will be introduced to the online course preoperatively
  Interventions: Behavioral: Wim Hof Method
- Standard Care Group (No Intervention): The control group will get the standard of care therapy after surgery.

INTERVENTIONS:
Behavioral: "Prepare for Surgery, Heal Faster" Program — This NYU program teaches patients how to feel calmer before surgery. Patients are taught relaxation techniques by phone or in person by trained NYU personnel. The program uses five steps to ease stress-related symptoms prior to surgery and improve help recovery time. By practicing deep relaxation, it is possible to reduce anxiety and promote a feeling of calmness. The patient swill be enrolled in the course preoperatively and will be ask to continue these meditations for ten weeks.
  Arms: Relaxation Group
Behavioral: Wim Hof Method — Patients will be enrolled in Wim Hof Method, a breathing/meditation program. This is a free online program, developed by a man named Wim Hof and his techniques. On this website, he explains the origins and methods behind his teachings ( https://www.wimhofmethod.com/iceman-wim-hof. ). Patients in this group will take the online free course provided by the Wim Hof Method. The patients will be introduced to the online course preoperatively. The three pillars of the WHM are 1) breathing/meditation, 2) stretching exercises and 3) gradual cold exposure. The patients will be told to concentrate on the breathing and meditation component, they may not be able to participate in the cold exposure (cold showers, ice baths) in the immediate post op period because of the open wounds.
  Arms: Meditation Group

SUMMARY:
Participants undergoing hand surgery will be assessed and compared for postoperative pain. The patients' experience of going through surgery will be evaluated. The patient satisfaction and patient assessed outcomes will be measured.

DETAILED DESCRIPTION:
Participants undergoing hand surgery will be randomized into either a control group or one of two groups that undergo mindfulness training during the perioperative period. One of the treatment groups will be enrolled in the program "Prepare for Surgery, Heal Faster" provided by NYU. The other treatment group will be enrolled in Wim Hof Method, a meditation program. This program is not provided by NYU, but instructions will be provided to the patient on how to complete the meditative exercises involved in this established method. Postop pain medication and pain scores will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patient seen in Dr. Paksima's office
* Scheduled for hand surgery
* Aged 18+
* Able to provide consent

Exclusion Criteria:

* Less than 18 years old
* Inability to consent
* Not fluent in English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Change of Measured Pain | Day 0, 2 weeks, 6 weeks, 3 months, 1 year
  Pain will be measured by the visual analog scale (VAS) scale, The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."

SECONDARY OUTCOMES:
Change in Mindfulness Score of MAAS scale | Day 0, 2 weeks, 6 weeks, 3 months, 1 year
  Mindfulness will be measured by the Mindful Attention Awareness (MAAS) Scale. The Mindful Attention Awareness Scale (MAAS) is a 15-item self-report survey that measures the tendency to be fully aware of one's experience in the present moment without distraction or forgetfulness. Participants indicate whether they frequently or infrequently experience each item using a 6-point Likert scale: 1 (Almost Always), 2 (Very Frequently), 3 (Somewhat Frequently), 4 (Somewhat Infrequently), 5 (Very Infrequently), and 6 (Almost Never). The scale was developed with the understanding that people likely have better conscious access to information about their tendency to be mindless rather than mindful. As a result, the total score for the MAAS is computed by reverse-scoring and then summing all items

CONTACTS AND LOCATIONS:
Overall Officials: Nader Paksima, Principal Investigator — NYU Langone Health
Locations (1):
- NYUSoM, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
their data will only be used for this study's outcome measures